CLINICAL TRIAL: NCT00696475
Title: A Randomized, Double-Blind, Placebo-Controlled Study Assessing the Efficacy and Safety of Diazoxide Choline in Non-Diabetic Hypertriglyceridemic Subjects
Brief Title: Diazoxide Choline in Hypertriglyceridemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Essentialis, Inc. (Industry)
Collaborators: Medpace, Inc. (Industry)
Responsible Party: Neil M Cowen, PhD/Chief Scientific Officer, Essentialis
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PC007
Record Dates: First submitted 2008-06-10; First posted 2008-06-12 (Estimated); Last update posted 2010-11-08 (Estimated); Status verified 2010-11

CONDITIONS: Hypertriglyceridemia
MeSH Terms: conditions — Hypertriglyceridemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): Diazoxide equivalent dose
  Interventions: Drug: Diazoxide choline
- 2 (Experimental): Diazoxide equivalent dose
  Interventions: Drug: Diazoxide choline
- 3 (Experimental): Diazoxide equivalent dose
  Interventions: Drug: Diazoxide choline
- 4 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Diazoxide choline
  Arms: 1
Drug: Diazoxide choline
  Arms: 2
Drug: Diazoxide choline
  Arms: 3
Drug: Placebo
  Arms: 4

SUMMARY:
Hypertriglyceridemia affects 30% of the population in the US. Very high level of triglycerides is a known risk factor for pancreatitis. In addition, studies have shown that hypertriglyceridemia is an independent risk factor for cardiovascular disease.

Diazoxide is a KATP channel opener. It has been approved by the FDA as an oral suspension for the treatment of hyperinsulinemic hypoglycemic conditions and as an IV solution for malignant hypertension. Preclinical and clinical studies suggest that diazoxide can be a potential therapeutic agent for hypertriglyceridemia.

Diazoxide choline is a novel, highly crystalline proprietary salt of diazoxide, which has been formulated as a controlled-release tablet suitable for once per day dosing. This current study is designed to assess the effect of diazoxide choline on triglycerides in subjects with baseline hypertriglyceridemia. In addition, the effects on other lipid parameters, glucose and insulin, body weight as well as the safety and tolerability of diazoxide choline will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* triglycerides ≥ 250 mg/dL and < 600 mg/dL
* BMI between 18.5 and 45
* Signed informed consent form

Exclusion Criteria:

* Fasting glucose ≥ 126 mg/dL
* Glycosylated hemoglobin (HbA1c) > 6.5%
* LDL cholesterol > 190 mg/dL
* Known history of type I and II DM
* Known history of type I and III hyperlipidemia
* Weight change > 3 kg between screening and baseline visits
* Pregnancy or intention to become pregnant
* Presence of significant underlying conditions that may interfere with the assessments of the study drug

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2008-06; Primary Completion 2009-01 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
To assess the effect on triglycerides of repeated doses of Diazoxide Choline Controlled-Release Tablet over a period of 56 days in hypertriglyceridemic subjects | 8 weeks

SECONDARY OUTCOMES:
To assess the effect on other lipid parameters (LDL, HDL, VLDL, and non-HDL cholesterol), insulin, glucose and weight of repeated doses of Diazoxide Choline Controlled-Release Tablet over a period of 56 days in hypertriglyceridemic subjects | 8 weeks
To assess the safety and tolerability of repeated doses of Diazoxide Choline Controlled-Release Tablet over a period of 56 days in hypertriglyceridemic subjects | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Harold Bays, MD, Principal Investigator — L-MARC Research Center; Alan Forker, MD, Principal Investigator — St. Luke's Lipid and Diabetes Research Center; Cynthia Huffman, MD, Principal Investigator — Meridien Research; Michael Koren, MD, Principal Investigator — Jacksonville Center For Clinical Research; Andrew Lewin, MD, Principal Investigator — National Research Institute; Thomas Littlejohn, MD, Principal Investigator — Piedmont Medical Research Associates; David Morin, MD, Principal Investigator — TriCities Medical Research; Eli Roth, MD, Principal Investigator — Sterling Research Group, Ltd; Evan Stein, MD, Principal Investigator — Metabolic and Atherosclerosis Research Center (MARC); Philip Toth, MD, Principal Investigator — Midwest Institute for Clinical Research; Craig Thompson, MD, Principal Investigator — Frederick C. Smith Clinic; Glibert Weiner, MD, Principal Investigator — Allied Research International/Cetero Research
Locations (12):
- United States (12):
  - National Research Institute, Los Angeles, California
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Allied Research International/Cetero Research, Miami Gardens, Florida
  - Meridien Research, Tampa, Florida
  - Midwest Institute for Clinical Research, Indianapolis, Indiana
  - L-MARC Research Center, Louisville, Kentucky
  - St. Luke's Lipid and Diabetes Research Center, Kansas City, Missouri
  - Piedmont Medical Research Associates, Winston-Salem, North Carolina
  - Metabolic and Atherosclerosis Research Center (MARC), Cincinnati, Ohio
  - Sterling Research Group, Ltd, Cincinnati, Ohio
  - Frederick C. Smith Clinic, Marion, Ohio
  - TriCities Medical Research, Bristol, Tennessee